CLINICAL TRIAL: NCT02143063
Title: Extending Long-term Outcomes Through an Adaptive Aftercare Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sheila Alessi, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-090H-2; P50DA009241 (NIH)
Record Dates: First submitted 2014-02-24; First posted 2014-05-20 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Cocaine Use Disorder; Contingency Management
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard care (Active Comparator): standard care
  Interventions: Behavioral: standard care
- standard care plus traditional contingency managment (Active Comparator): prize contingency management on a traditional twice weekly schedule for cocaine abstinence
  Interventions: Behavioral: prize contingency management on a traditional twice weekly schedule for cocaine abstinence; Behavioral: standard care
- standard care plus variable interval contingency management (Experimental): prize contingency management on a variable interval schedule for cocaine abstinence
  Interventions: Behavioral: prize contingency management on a variable interval schedule for cocaine abstinence; Behavioral: standard care

INTERVENTIONS:
Behavioral: prize contingency management on a traditional twice weekly schedule for cocaine abstinence
  Arms: standard care plus traditional contingency managment
Behavioral: prize contingency management on a variable interval schedule for cocaine abstinence
  Arms: standard care plus variable interval contingency management
Behavioral: standard care

SUMMARY:
Reinforcement interventions have pronounced effects on reducing cocaine use. This study will evaluate a novel approach in which reinforcement frequency varies by patient performance. To test efficacy, 280 patients with cocaine use disorder will be randomly assigned to: standard care, standard care plus traditional twice weekly reinforcement, or standard care plus adaptive variable interval reinforcement.

DETAILED DESCRIPTION:
Reinforcement interventions have pronounced effects on reducing cocaine use. We developed and evaluated a low-cost reinforcement intervention, systematically moving it through the Stages of development to dissemination and broad clinical implementation. In an ongoing project, reinforcement interventions are yielding benefits when reinforcers are provided at treatment initiation and for longer durations. However, less than half of patients remain engaged for 12 weeks with traditional reinforcement interventions, which require frequent attendance for monitoring and reinforcing abstinence. Interventions that extend into aftercare and that are acceptable to and efficacious in preventing long-term relapse are critically needed.

Reinforcement interventions are efficacious during periods they are in effect, and pilot data show that variable interval (VI) reinforcement schedules, once behavior change occurs, hold potential for maintaining gains when administered infrequently. Assessing methods to extend benefits of these interventions is of paramount scientific and clinical concern. This study will evaluate a novel approach in which reinforcement frequency varies by patient performance. In this intervention, reinforcement will be available for 24 weeks, on a progressive VI schedule, that adapts according to patient status. Patients who maintain abstinence earn maximum reinforcers as infrequently as every three weeks on average, while frequency of monitoring and reinforcing abstinence will increase in those who relapse until abstinence is re-instated.

To test efficacy, 280 patients with cocaine use disorder will be randomly assigned to: standard care (SC), SC+traditional twice weekly reinforcement, or SC+adaptive VI reinforcement. Evaluations will be completed at baseline and throughout 18 months to assess objective and self-reported indices of drug use, psychosocial problems, and HIV risk behaviors. Primary hypotheses are (1) the adaptive VI reinforcement intervention will improve outcomes relative to standard care during the treatment period and throughout follow-up, and (2) the adaptive VI reinforcement intervention will improve outcomes relative to the traditional reinforcement system. This study will also evaluate the roles of cognitive control and treatment outcome. Patients with better cognitive control are expected to maintain longer durations of abstinence across conditions. If these measures differentially relate to outcomes across treatments, such results suggest the potential of pairing reinforcement interventions to individuals most likely to benefit from them; they may also indicate possible markers of response in a treatment-specific manner. If cognitive indices mediate treatment response, future studies can refine interventions to improve cognitive processes and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* be age 18 years or older
* have a cocaine use disorder diagnosis
* be willing to sign informed consent and able to pass an informed consent quiz

Exclusion Criteria:

* serious, uncontrolled psychiatric illness
* in recovery from pathological gambling
* do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Petry, Ph.D., Principal Investigator — UConn Health
Locations (4):
- United States (4):
  - Regional Network of Programs, Inc., Bridgeport, Connecticut
  - Alcohol and Drug Recovery Centers, Inc., Hartford, Connecticut
  - The Hospital of Central Connecticut at New Britain General, New Britain, Connecticut
  - Behavioral Health Network, Inc., Springfield, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care (SC): Standard care IOP treatment for cocaine use disorder. In addition, SC participants submitted urine samples during the 24-week intervention phase. Patients selected two days a week on which drug screens might occur (e.g., M/Th, T/F). On the morning of each potential drug screen day, research staff texted participants to indicate if a sample was due. In weeks 1-3, urine screens occurred on two days per week. In weeks 4-9, screens occurred on one randomly selected day each week. In weeks 10-24, drug screens occurred once every 2-3 weeks on average. After a missed sample, the next two screen days were prompted for sample submission. An algorithm developed in-house was used to generate and monitor the drug screen schedule. Participants received $2 per requested sample submitted plus a $20 bonus for submitting all requested samples in a 4-week period. The goal was to result in 18 samples on average, equivalent relative to the new SC plus variable interval CM condition.
- Standard Care Plus Traditional Contingency Management: Standard care plus "standard" prize contingency management twice weekly for urine screens indicating cocaine abstinence. Urine screens occurred on the same monitoring schedule described for the SC condition, including $2 per requested sample submitted and a $20 bonus for all requested samples in a 4-week period. In addition, participants received chances for prizes on a escalating reinforcement schedule and with a reset condition for unexcused missed samples. Mean maximum earnings for cocaine-negative urine screens was $460 in prizes.
- Standard Care Plus Variable Interval Contingency Management: Standard care plus prize contingency management on a variable interval schedule for cocaine abstinence. Relative to the traditional CM condition, in this condition, the frequency of samples to earn reinforcement decreased over time contingent on achieving periods of sustained abstinence. The schedule was designed to result in an average of at least 18 urine samples over 24 weeks among participants maintaining abstinence. Participants received the sample compensation for submitted urine samples regardless of results as in the other two conditions.
Period: Overall Study
Arm/Group | Standard Care (SC) | Standard Care Plus Traditional Contingency Management | Standard Care Plus Variable Interval Contingency Management
Started | 61 | 105 | 108
Completed | 45 | 75 | 78
Not Completed | 16 | 30 | 30
Not completed — Lost to Follow-up | 16 | 28 | 29
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Death | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard Care Plus Traditional Contingency Managment: prize contingency management on a traditional twice weekly schedule for cocaine abstinence
  prize contingency management on a traditional twice weekly schedule for cocaine abstinence
  standard care
- Standard Care Plus Variable Interval Contingency Management: prize contingency management on a variable interval schedule for cocaine abstinence
  prize contingency management on a variable interval schedule for cocaine abstinence
  standard care
- Total: Total of all reporting groups
Arm/Group | Standard Care | Standard Care Plus Traditional Contingency Managment | Standard Care Plus Variable Interval Contingency Management | Total
Number analyzed (Participants) | 61 | 105 | 108 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (9.2) | 40.7 (9.6) | 39.7 (10.1) | 40.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 57 | 58 | 147
  Male | 29 | 48 | 50 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 23 | 27 | 64
  Not Hispanic or Latino | 47 | 81 | 81 | 209
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 35 | 30 | 81
  White | 33 | 52 | 64 | 149
  More than one race | 5 | 4 | 6 | 15
  Unknown or Not Reported | 6 | 12 | 8 | 26
Region of Enrollment [Number; unit: participants]
  United States | 61 | 105 | 108 | 274

OUTCOME MEASURES:

1. Primary Outcome: Longest Duration of Abstinence From Cocaine
Description: Longest duration of consecutive cocaine-negative urine toxicology tests
Time Frame: baseline through 6 months
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Standard Care | Standard Care Plus Traditional Contingency Managment | Standard Care Plus Variable Interval Contingency Management
Number analyzed (Participants) | 58 | 104 | 104
weeks | 4.14 [1.14 to 8.86] | 6.64 [2.79 to 13.57] | 6.93 [2.14 to 12.57]
Statistical Analysis 1: Comparison: Standard Care vs Standard Care Plus Variable Interval Contingency Management; Test type: Superiority; p = .01, Wilcoxon (Mann-Whitney); comparison of rank sum = 3752.0
Statistical Analysis 2: Comparison: Standard Care Plus Traditional Contingency Managment vs Standard Care Plus Variable Interval Contingency Management; Test type: Superiority; p = .78, Wilcoxon (Mann-Whitney); comparison of rank sum = 5287.5

2. Secondary Outcome: Longest Duration of Abstinence From All Substances Tested
Description: Based on breath and urine toxicology tests (alcohol, methamphetamine, cocaine, opioids, THC, amphetamine, benzodiazepines)
Time Frame: baseline through 6 months
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Standard Care | Standard Care Plus Traditional Contingency Managment | Standard Care Plus Variable Interval Contingency Management
Number analyzed (Participants) | 58 | 104 | 104
weeks | 4.75 [0.68 to 8.04] | 5.93 [1.57 to 12.64] | 5.71 [1.57 to 11.64]
Statistical Analysis 1: Comparison: Standard Care vs Standard Care Plus Traditional Contingency Managment; Primary Aim 1: Compare the standard care and standard care plus traditional CM conditions; Test type: Superiority; p = .02, Wilcoxon (Mann-Whitney); comparison of rank sum = 3675.5
Statistical Analysis 2: Comparison: Standard Care Plus Traditional Contingency Managment vs Standard Care Plus Variable Interval Contingency Management; Test type: Superiority; p = .61, Wilcoxon (Mann-Whitney); comparison of rank sum = 5189.5

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Standard Care | Standard Care Plus Traditional Contingency Managment | Standard Care Plus Variable Interval Contingency Management
All-Cause Mortality (participants affected / at risk) | 0/61 | 1/105 | 1/108
Serious Adverse Events (participants affected / at risk) | 46/61 | 66/105 | 77/108
Other Adverse Events (participants affected / at risk) | 12/61 | 7/105 | 9/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=61) | Standard Care Plus Traditional Contingency Managment (N=105) | Standard Care Plus Variable Interval Contingency Management (N=108)
Inpatient substance use treatment (Social circumstances) | 27 (58) | 40 (59) | 47 (66)
Inpatient psychiatric treatment (Psychiatric disorders) | 9 (18) | 5 (7) | 12 (16)
Inpatient medical treatment (General disorders) | 12 (19) | 20 (28) | 18 (25)
Death (General disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=61) | Standard Care Plus Traditional Contingency Managment (N=105) | Standard Care Plus Variable Interval Contingency Management (N=108)
Suicidal Ideation (Psychiatric disorders) | 9 (11) | 4 (5) | 6 (6)
ER visit for overdose (General disorders) | 3 (3) | 3 (5) | 3 (3)

LIMITATIONS AND CAVEATS:
Analyses presented assessed outcomes at the group-level and using main a priori analytic methods. Additional analyses should assess outcomes in the context of potential baseline predictors, assess for patterns in individual-level trajectories over time and by group, and incorporate additional advanced analytic techniques.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT02143063/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT02143063/ICF_001.pdf